CLINICAL TRIAL: NCT03477812
Title: Sleep and Nocturnal Enuresis: Ambulatory Polysomnographic Study at Home - Differences Between Monosymptomatic Nocturnal Enuresis Patients and Healthy Controls
Brief Title: Sleep and Nocturnal Enuresis: Ambulatory Polysomnographic Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: Sleep and nocturnal enuresis
Record Dates: First submitted 2018-02-05; First posted 2018-03-26 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-01

CONDITIONS: Nocturnal Enuresis; Polysomnography
MeSH Terms: conditions — Nocturnal Enuresis | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy children: Healthy children 7-14 years of age.
  Interventions: Device: Polysomnography (Full sleep registration)
- Nocturnal enuresis with polyuria: Children with nocturnal enuresis and polyuria aged 7-14 years.
  Interventions: Device: Polysomnography (Full sleep registration)
- Nocturnal enuresis without polyuria: Children without nocturnal enuresis and polyuria aged 7-14 years.
  Interventions: Device: Polysomnography (Full sleep registration)

INTERVENTIONS:
Device: Polysomnography (Full sleep registration) — For the healthy children two nights of polysomnography. For the children with nocturnal enuresis one night of polysomnography.

SUMMARY:
Full ambulatory polysomnography at home performed two nights in 30 healthy children and one night in 30 children with mono-symptomatic nocturnal enuresis (15 with polyuria and 15 without polyuria). The children will be aged 7-14 years of age.

The sleep will be evaluated on sleep quality, number of periodic limb movements per hour, blood pressure and pulse, beat to beat variation by electrocardiography during sleep, respiration during sleep, nocturnal urine production, and enuresis episodes.

DETAILED DESCRIPTION:
Purpose and perspectives:

The purpose of the study is to investigate the quality of sleep, the sleep architecture and the intra-individual variation from night to night in healthy children and children with mono-symptomatic nocturnal enuresis (MNE) using full polysomnography at home.

Hypotheses:

* There is large intra-individual night to night variation in sleep quality and architecture.
* Children with MNE have different sleep architecture than healthy children when looking at sleep quality and arousals.
* Periodic limp movements at sleep is more frequent in children with MNE than in healthy children.

Design:

The study is a case-control study.

Materials and methods:

The study will recruit 30 healthy children and 30 children with MNE (15 with polyuria and 15 without polyuria) recruited from the Childrens Incontinence Center at the Department of Pediatrics and Adolescent Medicine at Aarhus University Hospital. Children of both sexes aged between 7 and 14 years of age will be enrolled. Children and their parents will be informed about the study both verbally and in written. Written informed consent from both parents must be obtained before the children can be enrolled in the study.

The healthy children will go through two nights of full polysomnography to be able to view intra-individual changes. The children with MNE will only have to do one night of polysomnography.

Primary parameters:

* Sleep quality
* Number of periodic limb movements per hour
* Blood pressure and pulse
* Beat to beat variation by electrocardiography during sleep
* Respiration during sleep
* Nocturnal urine production
* Enuresis episodes

ELIGIBILITY:
Inclusion Criteria:

* 7-14 years of age
* Normal objective evaluation including blood pressure
* For healthy controls achieved continence both day and night before the age of 5.
* For children with nocturnal enuresis at least 3 wet nights per week.
* For children with enuresis clinical characteristics and at least one week of home recordings of nocturnal urine production and two days of full recording of fluid intake and urine production.

Exclusion Criteria:

* Obstipation (according to ROM IV criteria)
* Day incontinence or severe urgency
* Insomnia or known sleep disorders such as sleep walking, heavy snoring, night terrors or abnormal circadian rhythm.
* Present or former deceases in the urinary tract, liver or in the endocrinological system.
* Hypertension
* Treatment with medication at the time of the study
* ADHD, autism or other psychiatric disorders.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population will be 30 children with mono-symptomatic nocturnal enuresis aged from 7-14 years. The group of children with nocturnal enuresis will be split in two with 15 patients with polyuria and 15 without polyuria. The control group will be 30 healthy children aged 7-14 years of age.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-01-22 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Sleep efficiency | One night of polysomnography.
  Sleep efficiency will be calculated as the ratio of the total time spent asleep to the total time spent in bed

SECONDARY OUTCOMES:
Periodic limb movements during sleep | One night of polysomnography.
  Number of periodic limb movements per hour at sleep compared between the three groups.
Nocturnal urine production | One night of polysomnography.
  We will compare the nocturnal urine production in millilitres in the three groups.
Enuresis episodes | One night of polysomnography
  We are going to look at the time of the enuresis episode and compare it to the polysomnographic findings at that time.
Respiratory events during sleep | One night of polysomnography
  Respiration during sleep comparison between the three groups. This includes saturation, nasal air flow and movement of the stomach and chest. Together showing the number of respiratory events (apneas/hour).
Incidence of sleep disturbances | One night of polysomnography
  Percentage of children with clinical sleep disturbances between patients and controls
Intra-individual differences in sleep efficiency from night to night in healthy controls. | Two nights of polysomnography. Each evaluated after completing the two nights.
  Sleep efficiency (in percent) will be compared between the two nights of polysomnography in the healthy controls.
Intra-individual differences in periodic limb movements during sleep from night to night in healthy controls. | Two nights of polysomnography. Each evaluated after completing the two nights.
  Periodic limb movements during sleep will be compared between the two nights of polysomnography in the healthy controls.
Intra-individual differences in nocturnal urine production from night to night in healthy controls. | Two nights of polysomnography. Each evaluated after completing the two nights.
  Nocturnal urine production will be compared between the two study nights in the healthy controls.
Intra-individual differences in respiratory events from night to night in healthy controls. | Two nights of polysomnography. Each evaluated after completing the two nights.
  The number and kinds of respiratory events will be compared between the two study nights in the healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Søren Rittig, Professor, Study Chair — Aarhus University Hospital
Locations (1):
- Department of Pediatrics and Adolescent Medicine, Aarhus University Hospital, Aarhus, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No
Individual participant data is not going to be available to other researchers.

REFERENCES:
- [Derived] Pedersen MJ, Leonthin H, Mahler B, Rittig S, Jennum PJ, Kamperis K. Two nights of home polysomnography in healthy 7-14-year-old children - Feasibility and intraindividual variability. Sleep Med. 2023 Jan;101:87-92. doi: 10.1016/j.sleep.2022.10.027. Epub 2022 Oct 30. PMID 36368073